CLINICAL TRIAL: NCT00514748
Title: A Bilateral Interconnected DIEP Flap Based on One Vessel Pedicle for Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Yilin Cao, Plastic Surgery Hospital of Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 621125-2
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Mammaplasty
Keywords: breast reconstruction; DIEP; vessel pedicle
MeSH Terms: interventions — diclofenac hydroxyethylpyrrolidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients who receive breast reconstruction with bilateral DIEP flap based on bilateral vessel pedicles
  Interventions: Procedure: DIEP
- 2 (Experimental): Patient who receive breast reconstruction with vessel interconnected DIEP flap based on one vessel pedicle
  Interventions: Procedure: Interconnected DIEP

INTERVENTIONS:
Procedure: DIEP — flap survival, operation time, flap complications, donor site morbidity.
  Arms: 1
Procedure: Interconnected DIEP — flap survival, operation time, flap complications, donor site morbidity.
  Arms: 2

SUMMARY:
Bilateral DIEP flap needs two groups of vessel pedicles. We suppose that the bilateral DIEP flap may survive on one vessel pedicle by means of interconnection of bilateral DIEA. This study is aimed to build a interconnected vessel system of bilateral DIEP flap based on one vessel pedicle and observe its survival in breast reconstruction.

DETAILED DESCRIPTION:
The DIEP flap have become the most common and primary choice in autogenous tissue breast reconstruction nowadays. In cases with inadequate abdominal soft-tissue volume or abdominal midline scar, the bilateral DIEP flap is needed.However, it need two groups of recipient vessels. So it is unavailable in cases short of two groups of recipient vessels after radiotherapy. This study is aimed to solve the problems by interconnecting one of the branches of DIEA each side. The MDCT will be used to predict the branches and perforators of DIEA both sides. According to the branches of DIEAs, one branch will be anastomosed with that on contralateral side with only one vessel pedicle preserved on one side. We believe that the whole flap can be completely nourished with only one vessel pedicle by means of vessel interconnection.

ELIGIBILITY:
Inclusion Criteria:

* Breast lost after mastectomy
* With good general condition
* No pregnancy demand
* With additional soft tissue needed for reconstruction

Exclusion Criteria:

* With bad general condition
* DIEA damaged by previous surgery
* Limited abdominal tissue

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
the whole flap may survived on the single vessel pedicle. | more than one year after srugery

CONTACTS AND LOCATIONS:
Overall Officials: Jie Luan, MD, Study Chair — Plastic Surgery Hospital Affilicated to Chinese Academy of Medical Science
Locations (1):
- Plastic Surgery Hospital, Beijing, China

REFERENCES:
- [Background] Bains RD, Stanley PR, Riaz M. Avoiding donor-site complications with bilateral DIEP flaps in patients with subcostal scars. Plast Reconstr Surg. 2007 Jun;119(7):2337-2339. doi: 10.1097/01.prs.0000261064.22785.74. No abstract available. PMID 17519766
- [Background] Bains RD, Riaz M, Stanley P. Bilateral free DIEP breast reconstruction using contralateral internal mammary and ipsilateral thoracodorsal vessels. Plast Reconstr Surg. 2007 Apr 1;119(4):1385-1386. doi: 10.1097/01.prs.0000255180.17788.8c. No abstract available. PMID 17496625
- [Background] Lasso JM, Sancho M, Campo V, Jimenez E, Perez Cano R. Epiperitoneal vessels: more resources to perform DIEP flaps. J Plast Reconstr Aesthet Surg. 2008 Jul;61(7):826-9. doi: 10.1016/j.bjps.2007.03.004. Epub 2007 Apr 18. PMID 17446150
- [Background] Schoeller T, Wechselberger G, Roger J, Hussl H, Huemer GM. Management of infraumbilical vertical scars in DIEP-flaps by crossover anastomosis. J Plast Reconstr Aesthet Surg. 2007;60(5):524-8. doi: 10.1016/j.bjps.2006.11.008. Epub 2007 Jan 22. PMID 17399662
- [Background] Das-Gupta R, Busic V, Begic A. Deep inferior epigastric perforator flap (DIEP) breast reconstruction in the presence of a midline vertical scar. J Plast Reconstr Aesthet Surg. 2006;59(6):675-6. doi: 10.1016/j.bjps.2005.07.003. No abstract available. PMID 16817262
- [Background] Holm C, Mayr M, Hofter E, Ninkovic M. Perfusion zones of the DIEP flap revisited: a clinical study. Plast Reconstr Surg. 2006 Jan;117(1):37-43. doi: 10.1097/01.prs.0000185867.84172.c0. PMID 16404245
- [Background] Gill PS, Hunt JP, Guerra AB, Dellacroce FJ, Sullivan SK, Boraski J, Metzinger SE, Dupin CL, Allen RJ. A 10-year retrospective review of 758 DIEP flaps for breast reconstruction. Plast Reconstr Surg. 2004 Apr 1;113(4):1153-60. doi: 10.1097/01.prs.0000110328.47206.50. PMID 15083015
- [Background] Garcia-Tutor E, Murillo J. The ideal patient for the first breast reconstruction using a diep flap. Plast Reconstr Surg. 2003 Feb;111(2):947-8. doi: 10.1097/00006534-200302000-00087. No abstract available. PMID 12560733
- [Background] Vesely J, Stupka I, Drazan L, Holusa P, Licata P, Corradini B. DIEP flap breast reconstruction--new experience. Acta Chir Plast. 2001;43(1):3-6. PMID 11370256
- [Background] Tran NV, Buchel EW, Convery PA. Microvascular complications of DIEP flaps. Plast Reconstr Surg. 2007 Apr 15;119(5):1397-1405. doi: 10.1097/01.prs.0000256045.71765.96. PMID 17415232
- [Background] Blondeel PN. One hundred free DIEP flap breast reconstructions: a personal experience. Br J Plast Surg. 1999 Mar;52(2):104-11. doi: 10.1054/bjps.1998.3033. PMID 10434888